CLINICAL TRIAL: NCT04802512
Title: Investigation of the Turkish Validity and Reliability of the Telehealth Usability Questionnaire (TUQ)
Brief Title: Turkish Version of Telehealth Usability Questionnaire (TUQ)
Status: Completed | Type: Observational
Sponsor: Irem Hüzmeli (Other)
Responsible Party: Sponsor-Investigator, Irem Hüzmeli, Phd lecturer, Mustafa Kemal University
Organization: Mustafa Kemal University (Other)
Other Study IDs: HatayMustafaKU
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Health Care Acceptor; Health Knowledge, Attitudes, Practice; Patient Participation
MeSH Terms: conditions — Patient Acceptance of Health Care; Behavior; Patient Participation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: patients who were used telehealth
  Interventions: Procedure: validity and reability study
- health professional: health professional who were used telehealth.
  Interventions: Procedure: validity and reability study

INTERVENTIONS:
Procedure: validity and reability study — validity and reliability assessment of the Turkish version of the Telehealth Usability Questionnaire (TUQ)

SUMMARY:
The Telehealth Usability Questionnaire (TUQ) was developed to evaluate the usability of telehealth applications and services. The Turkish validity and reliability study of the scale, originally in English, has not been conducted before.

The aim of this study is to develop the Turkish version of the Telehealth Usability Questionnaire (TUQ), which is a new stability tool, and to report its reliability assessment.

DETAILED DESCRIPTION:
The Telehealth Usability Questionnaire (TUQ) turkish version will be asked by using google forms to participants whom use telehealth.

ELIGIBILITY:
Inclusion Criteria:

Participants will undergo screening to confirm eligibility, completion of initial screening form, and MMSE evaluation. Study subjects were enrolled with MMSE scores between 29-30, inclusive (healthy/control), 25-28, inclusive (mild cognitive impairment), and 10-24 (dementia).

-

Exclusion Criteria:

* Unable to complete computerized and standard pencil-and-paper based assessments

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Turkish validity and reliability of the scale, which was created to evaluate the usability of the telehealth service for service users (patients) and providers (health professional), will be investigated.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2022-06-12 (Actual)

PRIMARY OUTCOMES:
Reliability and Validity of TUQ by Correlation Analysis. | 12 month
  with telehealth will be researched

CONTACTS AND LOCATIONS:
Overall Officials: Irem Huzmeli, Phd, Study Director — Mustafa Kemal University; Esra Dogru Huzmeli, Assoc Prof., Principal Investigator — Mustafa Kemal University; Mehmet Karadağ, Asist. Prof., Study Chair — Mustafa Kemal University
Locations (2):
- Turkey (Türkiye) (2):
  - Hatay Mustafa Kemal University, Hatay, Merkez
  - Online, Hatay

IPD SHARING:
Plan to Share IPD: Undecided